CLINICAL TRIAL: NCT02174835
Title: A Phase 1, Single-center, Randomized, Open-label Study to Assess the Pharmacokinetics, Safety and Tolerability of AVP-786 (Deuterated [d6] Dextromethorphan Hydrobromide/Quinidine Sulfate) in Healthy Volunteers
Brief Title: A Phase-1 Study to Assess the Pharmacokinetics, Safety and Tolerability of AVP-786 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avanir Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 13-AVR-134
Record Dates: First submitted 2014-06-23; First posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Healthy Volunteers; deuterated dextromethorphan; deuterated dextromethorphan with quinidine
MeSH Terms: interventions — dextromethorphan - quinidine combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort A - Period 1 (Experimental): Twice daily dosing orally for 7 days
  Interventions: Drug: AVP-786
- Cohort A - Period 2 (Active Comparator): Twice daily dosing orally for 7 days
  Interventions: Drug: AVP-923
- Cohort A - Period 3 (Experimental): Twice daily dosing orally for 7 days
  Interventions: Drug: AVP-786
- Cohort B - Period 1 (Experimental): Twice daily dosing orally for 7 days
  Interventions: Drug: AVP-786
- Cohort B - Period 2 (Active Comparator): Twice daily dosing orally for 7 days
  Interventions: Drug: AVP-923
- Cohort B - Period 3 (Experimental): Twice daily dosing orally for 7 days
  Interventions: Drug: AVP-786

INTERVENTIONS:
Drug: AVP-786
  Arms: Cohort A - Period 1; Cohort A - Period 3; Cohort B - Period 1; Cohort B - Period 3
Drug: AVP-923
  Arms: Cohort A - Period 2; Cohort B - Period 2

SUMMARY:
To assess the multiple-dose pharmacokinetics (PK), safety and tolerability of AVP-786 (deuterated [d6] dextromethorphan hydrobromide [DM]/quinidine sulfate [Q]) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males
* 18 - 45 years of age
* BMI 18 - 30 kg/m2

Exclusion Criteria:

* History or presence of significant disease
* History of substance abuse and/or alcohol abuse with the past 3 years
* Use of tobacco-containing or nicotine-containing products within 6 months
* Use of any prescription or the over-the-counter medications within 14 days

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of AVP-786 | 7 days

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) for AVP-786 | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Sepehr Shakib, M.D., Principal Investigator — CMAX
Locations (1):
- CMAX, Adelaide, South Australia, Australia